CLINICAL TRIAL: NCT03196986
Title: Efficacy and Safety of First-line mil60 Plus Paclitaxel/Carboplatin Versus Bevacizumab Plus Paclitaxel/Carboplatin in Patients With Advanced and Recurrent Non-squamous Non-small Cell Lung Cancer: a Randomized, Double-blind, Phase 3 Study
Brief Title: mil60 Versus Bevacizumab in Patients With Treatment-naïve Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: mil60-CT02
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mil60 (Experimental): mil60 (15mg/kg) was co-administered intravenously with 4 to 6-cycle paclitaxel/carboplatin, non-progressive patients are then given with maintenance single-agent mil60 (7.5mg/kg) until disease progression, intolerable toxicity, or withdrawal.
  Interventions: Drug: mil60
- Bevacizumab (Active Comparator): Bevacizumab (15mg/kg) was co-administered intravenously with 4 to 6-cycle paclitaxel/carboplatin, non-progressive patients are then given with maintenance single-agent mil60 (7.5mg/kg) until disease progression, intolerable toxicity, or withdrawal.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: mil60 — 15mg/kg in combination with paclitaxel/carboplatin for 6 cycles, then maintains at 7.5mg/kg
  Other Names: No other intervention name
  Arms: mil60
Drug: Bevacizumab — 15mg/kg in combination with paclitaxel/carboplatin for 6 cycles, then switched to mil60 at 7.5mg/kg
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
This randomized, double-blind, multi-center phase 3 study is aimed to compare the efficacy and safety of mil60 with bevacizumab as first-line treatment when combined with standard chemotherapy (paclitaxel/carboplatin) in treatment-naive patients with advanced or recurrent non-squamous NSCLC.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, parallel-group Phase 3 clinical trial evaluating the efficacy and safety of mil60 plus paclitaxel and carboplatin versus bevacizumab plus paclitaxel and carboplatin in first-line treatment for patients with advanced (unresectable, locally advanced, recurrent or metastatic) non-squamous NSCLC.The primary objective of the study was to compare the Objective Response Rate according to RECIST 1.1 of mil60 in combination with paclitaxel plus carboplatin and bevacizumab plus paclitaxel plus carboplatin in the treatment of advanced or recurrent non-squamous NSCLC subjects.

ELIGIBILITY:
Inclusion Criteria:

* signed inform consent form(ICF)
* Aged 18-75 years, male or female
* Histologically or cytologically documented inoperable, local advanced (stage IIIB), metastatic (stage IV), or recurrent non-squamous NSCLC
* At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Patients of childbearing potential must agree to use effective contraceptive measures during study treatment and for 6 months after receiving last study treatment

Exclusion Criteria:

* Mixed non-small cell lung cancer with squamous cell carcinoma component, or small cell carcinoma
* Patients with known Anaplastic Lymphoma Kinase（ALK） or C-Ros Oncogene 1 Receptor Tyrosine Kinase （ROS1）rearrangement
* History of hemoptysis within 3 months prior to screening with blood volume more than 2.5 mL
* Evidence of tumor invading major blood vessels on imaging
* Patients with brain metastasis, spinal cord compression or carcinomatous meningitis history
* Uncontrolled hypertension, prior history of hypertensive crisis and hypertensive encephalopathy
* Clinically significant cardiovascular disease but not limited to active infections; unstable angina; stroke or transient cerebral ischemia; myocardial infarction; congestive heart-failure; serious cardiac arrhythmia, hepatic, renal or metabolic disease requiring medication during the study
* History of radical radiotherapy to the thorax within 6 months
* Serious, non-healing wound, active ulcer, or untreated bone fracture, or major surgical procedure within 28 days prior to randomization or anticipation of need for major surgery during the course of the study
* Recent or current treatment with aspirin or other non-steroidal anti-inflammatory drugs (NSAID) known to inhibit platelet function within 10 days prior to first dose of study treatment
* Recent or current treatment with anticoagulants or thrombolytic agent within 10 days prior to first dose of study treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Percentage of patients with complete remission or partial response

SECONDARY OUTCOMES:
Objective response rate | 26 months
  Percentage of patients with complete remission or partial response
Duration of response | 24 months
  Interval from the onset of a complete remission or partial response until evidence of disease progression or death
Progression-free survival | 24 months
  Interval between randomization and disease progression or death
Disease control rate | 24 months
  Percentage of patients with complete remission, partial response and stable disease
Overall survival | 30 months
  the time from randomisation to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Institute/Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Shenzhen Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wan R, Dong X, Chen Q, Yu Y, Yang S, Zhang X, Zhang G, Pan Y, Sun S, Zhou C, Hong W, Zhao H, Yang L, Huang L, Wu R, Zang A, Ma R, Wu L, Lv D, Fu X, Han J, Li W, Duan J, Wang K, Jiang O, Chen Y, Guo Z, Gao H, Wen J, Wang S, Zhao E, Li G, Yue L, Liang L, Zeng A, Wang X, Zhu Y, Pan H, Dai Z, Feng W, Zhao G, Lin C, Li C, Li N, Bao Y, Li Y, Su Y, Zhao M, Fang H, Zhu Y, Zhang Y, Ding L, Wang Y, Yuan X, Wang J. Efficacy and safety of MIL60 compared with bevacizumab in advanced or recurrent non-squamous non-small cell lung cancer: a phase 3 randomized, double-blind study. EClinicalMedicine. 2021 Nov 19;42:101187. doi: 10.1016/j.eclinm.2021.101187. eCollection 2021 Dec. PMID 34841235